CLINICAL TRIAL: NCT06489834
Title: Group Drumming for Improving the Health of Community-Dwelling Elderly
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Lions Befriender (Unknown); Toteboard (Unknown); Institute of Mental Health, Singapore (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: 2023-2642
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Quality of Life; Depression; Sleep; Blood Pressure; Grip
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Waitlist control group study with control group undergoing intervention 8 weeks after intervention group has ceased
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor would be blinded to which arm the participants is in. Investigator will also be blinded to the treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drumming Arm (Active Comparator): Participants in this arm will undergo weekly group drumming for 8 weeks.
  Interventions: Other: Group Drumming
- Waitlist Control Arm (No Intervention): Participants in this arm will not undergo any intervention while the intervention arm is ongoing and assessed for comparison.

INTERVENTIONS:
Other: Group Drumming — Weekly group drumming for 8 weeks
  Arms: Drumming Arm

SUMMARY:
The study seeks to examine the effects that recreational group drumming has on the health of the community- dwelling elderly. It is hypothesized that it has positive and sustainable effects on various health outcome measures.

DETAILED DESCRIPTION:
The study seeks to examine the effects that recreational group drumming has on the health of the community- dwelling elderly. It is hypothesized that it has positive and sustainable effects on various health outcome measures.

One of the primary outcome measure is the quality of life of the participants, which will be measured using the European Quality of Life-5 Dimensions (EQ5D). It is a measure of health status from the EuroQoL. Group primarily designed for self-completion by respondents and is validated locally. The score ranges from 0 (death) to 1 (full health), with 5 dimensions comprising of mobility, self-care, usual activities, pain/discomfort and anxiety/ depression.

The other primary outcome measures include:

i. The Geriatric Depression Scale (GDS), which is a tool used for elderly population to evaluate the level of depressive symptoms of an individual over the past week, has been validated locally. It is a self-reported questionnaire consisting of 15 items. Maximum score of 15 and minimum of 0. Score equal or greater than 6 out of 15 is considered to be indicator of depression.

ii. The Pittsburgh Sleep Quality Index (PSQI) is a self-reported measure of sleep quality. It is a 19-item scale grouped into 7 equally weighted component scores. The global score ranges from 0 to 21, with poorer sleep quality indicated by a higher global score.

iii. (Social Effects) The Lubben Social Network Scale (LSNS) is a self-reported measure designed to gauge social isolation in the elderly. It measures frequency, size and closeness of contacts for the participant's social network by assessing the participant's perceived level of support received from friends and families.

The secondary outcomes are broadly categorized into psychological effects, social effects, and physical effects as listed below:

1. Psychological Effects The Mini Mental State Examination (MMSE) is a commonly used screening tool for cognitive impairment worldwide. A score of less than 25 out of maximum of 30 is often suggestive of an underlying cognitive impairment.
2. Physical Effects

   i. Resting blood pressure and heart rate

ii. Grip strength - popular indicator of physical functioning

iii. Minnesota Manual Dexterity Test

It is hypothesized that recreational group drumming has positive and sustainable effects on various health outcome measures.

The research study will be conducted in two phases. Phase 1 is the randomized controlled study comparing the intervention with independent concurrent controls. Phase 2 will involve providing the intervention to the control subjects from phase 1, where subjects act as their own controls pre to post intervention.

Each drumming session would have 20 participants, excluding two facilitators. This 'Bridging Rhythm with Wellness Programme' will be organised by Lions Befrienders Singapore. These drumming sessions will be held in the Active Ageing Centres (AACs) under Lions Befirenders.

Recruited study participants will be issued Study ID upon enrolment into study. Phase 1 Phase 1 is a randomized controlled trial with a planned ratio of participants of 1:1 in the intervention group (Group A) and control group (Group B). Unlike the pilot study, a crossover will not be conducted in view of (i) difficulties in quantifying a sufficient washout period for such an intervention and (ii) a possible learned effect being carried over.

Participants will be recruited from senior activity centre and randomized into either group within their respective senior activity centre.

All participants in phase 1, be it those randomised into control or intervention group, will be subjected to the following study procedures.

Clinical and patient related outcome data will be collected at the participants' respective senior activity centres at 4 time points:

1. At the start of the study
2. Midpoint of intervention (Week 4)
3. Completion of intervention (Week 8)
4. 4 Weeks post-intervention (Week 12) For assessments done at first study timepoint (i.e. start of study assessments), it can be completed 2-3 weeks prior to commencement of each centre's drumming session. This is to allow study team members to have time to complete the required baseline assessments prior to commencement of study intervention.

All study assessments to be completed within study timepoint week with 3 working date window period before and after study timepoint week.

Participants will be asked to complete the following questionnaires and clinical tests:

1. European Quality of Life-5 Dimensions (EQ5D)
2. Geriatric Depression Scale (GDS)
3. Pittsburgh Sleep Quality Index (PSQI)
4. Mini Mental State Examination (MMSE)
5. Lubben Social Network Scale (LSNS)
6. Katz ADL
7. Blood Pressure
8. Heart Rate
9. Grip Strength with Dynamometer
10. Minnesota Manual Dexterity Test
11. Study Data Collection Form Study participants may be contacted via phone calls to complete required questionnaires. Participants will be provided a research letter if any incidental finding have been found.

Phase 2 In phase 2, subjects in Group B or control group in phase 1, will be offered the opportunity to undergo the intervention at least 4 weeks after the intervention group has concluded Phase 1. Being control subjects in phase 1, these subjects have the baseline values for various measures accurately established prior to intervention. These subjects will act as their own controls, and the effect of the intervention will be assessed by comparing the post treatment values against the baseline measures prior to intervention.

Similar outcome measures will be measured at the time points relative to the baseline measurements, for both phase 1 and phase 2 studies.

Subjects (Group A of phase 1 and subjects of phase 2) will undergo a group drumming course under the Bridging Rhythm with Wellness Programme, comprising of 8 weekly sessions that last for an hour each. Participants cannot be blinded in the study as whoever playing instruments will be aware of the intervention. To protect against contamination, participants of the two groups will be assessed at different times.

In this group drumming course, a variety of percussion instruments will be used inn these sessions, including the conga, cowbell, Djembe, Ashiko, Tan-tans, Dunun, shakers and wood blocks. These instruments will be rotated among the participants from session to session. Participants will be seated comfortably in a circle on chairs within their assigned group, and the percussion instrument will be placed in front of them within reach. Each session will be led by 2 experienced artist-facilitators skilled in leading group drumming courses (1 fixed main facilitator, 1 co-facilitator). The artist-facilitators will be blinded to the participants' backgrounds, psychological and physical health profiles. Artist-facilitators will encourage free play, expression and interaction amongst participants through playing of instruments.

ELIGIBILITY:
Inclusion Criteria:

Individuals who are:

* Aged 60 years old and above (by year of age)
* Able to understand English and/or Mandarin, and
* Able to engage in the group drumming activity conducted (e.g. capable of light exercises while seated)

Exclusion Criteria:

Individuals who are:

* On palliative care, and/or
* Bed-bound
* Have severe hearing impairment such that they are unable to engage in group drumming sessions

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 12 weeks
  European Quality of Life-5 Dimensions (EQ5D) Will be measured. The score ranges from 0 (death) to 1 (full health), with 5 dimensions comprising of mobility, self-care, usual activities, pain/discomfort and anxiety/ depression.
Depression | 12 weeks
  Geriatric Depression Scores will be measured. Scores will range from 0-15. Those will lower scores will have higher risk of depression
Sleep Quality | 12 weeks
  Pittsburg Sleep quality index will be used to measure this outcome

SECONDARY OUTCOMES:
Psychological effects | 12 weeks
  Mini Mental State Examination (MMSE)will be measured. A score of less than 25 out of maximum of 30 is often suggestive of an underlying cognitive impairment.
Resting Blood Pressure | 12 weeks
  Resting Blood pressure will be measured at baseline and at 12 weeks. Both systolic and diastolic pressure would be captured in mmHg
Heart Rate | 12 weeks
  Resting Heart Rate will be measured at baseline and at 12 weeks. This would be in beats/minute

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yap AF, Kwan YH, Tan CS, Ibrahim S, Ang SB. Rhythm-centred music making in community living elderly: a randomized pilot study. BMC Complement Altern Med. 2017 Jun 14;17(1):311. doi: 10.1186/s12906-017-1825-x. PMID 28615007
- [Background] Smith C, Viljoen JT, McGeachie L. African drumming: a holistic approach to reducing stress and improving health? J Cardiovasc Med (Hagerstown). 2014 Jun;15(6):441-6. doi: 10.2459/JCM.0000000000000046. PMID 24983262
- [Background] Miyazaki A, Okuyama T, Mori H, Sato K, Ichiki M, Nouchi R. Drum Communication Program Intervention in Older Adults With Cognitive Impairment and Dementia at Nursing Home: Preliminary Evidence From Pilot Randomized Controlled Trial. Front Aging Neurosci. 2020 Jul 2;12:142. doi: 10.3389/fnagi.2020.00142. eCollection 2020. PMID 32714176